CLINICAL TRIAL: NCT03469349
Title: A Randomized, International, Multicenter, Parallel Group, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Actovegin 12-Week Treatment Given First Intravenously and Subsequently Orally in Subjects With Peripheral Arterial Occlusive Disease Fontaine Stage IIB
Brief Title: Actovegin 12-Week Treatment Given First Intravenously and Subsequently Orally in Participants With Peripheral Arterial Occlusive Disease Fontaine Stage IIB
Acronym: APOLLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Actovegin-3001; 2017-004741-24 (EudraCT Number); U1111-1201-7990 (Other: WHO)
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Arterial Diseases
Keywords: Drug Therapy
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Actovegin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actovegin 1200 mg (Experimental): Actovegin 1200 milligram (mg), intravenously, once daily for up to 2 weeks followed by actovegin 200 mg, tablets, orally, thrice daily (TID) (1200 mg/day) for up to 10 weeks.
  Interventions: Drug: Actovegin
- Placebo (Placebo Comparator): Actovegin placebo-matching, intravenously, once daily for up to 2 weeks and actovegin placebo-matching tablets, orally, TID for up to 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Actovegin — Actovegin intravenous infusion and tablets.
  Arms: Actovegin 1200 mg
Drug: Placebo — Actovegin placebo-matching intravenous infusion and tablets.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of actovegin in participants with peripheral arterial disease (PAD) Fontaine Stage IIB.

DETAILED DESCRIPTION:
The study will enroll approximately 366 participants. Participants will be randomly assigned to one of the two treatment groups in 1:1 ratio:

1. Actovegin
2. Placebo (dummy inactive substance) - this is a tablet/intravenous infusion that looks like the study drug but has no active ingredient

All participants will be asked to take intravenous infusion for 2 weeks followed by oral tablets for 10 weeks.

This multi-center trial will be conducted Russia, Georgia, and Kazakhstan. The overall time to participate in this study is 25 to 26 weeks. Participants will make multiple visits to the clinic, and 12 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a history of stable intermittent claudication lasting more than 6 months before Screening.
2. Has a diagnosis of peripheral arterial disease (PAD) (Code I70.2 according to the international classification of diseases-10th revision) Fontaine Stage IIB confirmed by ultrasound color duplex imaging.
3. Has a resting Doppler ankle-brachial index of less than or equal to (<=) 0.9.
4. Has intermittent claudication with initial claudication distance (ICD) less than (<) 200 meters.
5. Is not newly diagnosed with PAD and has a history of stable PAD therapy for at least 2 weeks before Screening.

Exclusion Criteria:

1. Has PAD Fontaine Stage III or IV (pain at rest, non-healing ulceration, or gangrene).
2. Has evidence of nonatherosclerotic PAD.
3. Has greater than (>) 25 percent (%) variability in absolute claudication distance (ACD) based on treadmill testing during the screening period.
4. Has lower extremity arterial reconstruction (surgical or endovascular) or sympathectomy within 3 months before Screening.
5. Is eligible for surgical/interventional reconstruction.
6. Had a myocardial infarction or major cardiac surgery within 3 months before Screening.
7. Has congestive heart failure (New York Heart Association Class III/IV).
8. Has uncontrolled diabetes mellitus (glycosylated hemoglobin [HbA1c >9%]) or diabetic polyneuropathy.
9. Has any other illness that significantly limits exercise capacity or other medical condition, including any psychiatric disorder that limits participation (in the judgement of the investigator).
10. The subject has received any prohibited medication within 14 days before Randomization (Day 1)
11. The subject is undergoing the supervised exercise training program by the time of Screening and is going to continue this program due to its effectiveness.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (20):
- Georgia (2):
  - Center of Vascular and Heart Disease, Tbilisi
  - Aversi Clinic, Tbilisi
- Kazakhstan (2):
  - "National scientific centre of oncology and transplantology", Astana
  - Regional Clinic Hospital, Shymkent
- Russia (16):
  - NSHI Road clinical hospital at Chelyabinsk station of OAO RZD, Chelyabinsk
  - Federal state budgetary research institution Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo
  - BMH Kursk regional clinical hospital of Healthcare department of Kursk region, Kursk
  - SBHI of Moscow city "City clinical hospital #29 n.a. N.E. Bauman of Moscow Healthcare department, Moscow
  - SBHI of Moscow healthcare department City clinical hospital #15 n.a. O.M Filatov of Moscow healthcare department, Moscow
  - SBHI of Moscow Research Institute of Emergency Medicine n.a. N.V. Sklifosofsky of Moscow Healthcare department, Moscow
  - Scientific Research Institute of Clinical and Experimental Lymphology - a branch of the Institute of Cytology and Genetics of the Siberian Branch of the Russian Academy of Sciences, Novosibirsk
  - BHI of Omsk region Regional clinical hospital, vessel surgery department, Omsk
  - FSBEI HE Rostov State Medical University of MoH of Russia, Rostov-on-Don
  - SBHI of Ryazan region Regional clinical cardiological dispensary, vessel surgery department/ FSBI of Ryazan Region "Ryazan State Medical Univesity n.a. I.P. Pavlov" of MoH of Russia, Ryazan
  - North-Western State Medical University named after I.I. Mechnikov, Saint Petersburg
  - SPb SBHI City multipurpose hospital #2, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Faculty surgery chair, cardio-vessel surgery department, Saint Petersburg
  - SPb SBHI Consulting and diagnostic center #85, Saint Petersburg
  - State Healthcare Institution of Saratov region "Region clinical hospitai", Saratov
  - Municipal State Budgetary Healthcare Institution of Sochi "City hospital 4", Sochi

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 19 investigative sites in Russia, Kazakhstan and Georgia from 01 May 2018 to 28 August 2019.
Pre-assignment Details: Participants with peripheral arterial occlusive disease (PAD) Fontaine stage IIB were enrolled in this study to receive either actovegin or placebo in a 1:1 ratio.
Groups:
- Placebo: Actovegin placebo-matching infusion, intravenously, once daily for up to 2 weeks followed by actovegin placebo-matching tablets, orally, thrice daily for up to 10 weeks.
- Actovegin 1200 mg: Actovegin 1200 milligram (mg), infusion, intravenously, once daily for up to 2 weeks followed by actovegin 200 mg, tablets, orally, thrice daily (1200 mg/day) for up to 10 weeks.
Period: Overall Study
Arm/Group | Placebo | Actovegin 1200 mg
Started | 182 | 184
Completed | 177 | 174
Not Completed | 5 | 10
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Progressive Disease | 0 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 2 | 4

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who were randomized and received at least 1 dose of double-blind study medication.
Groups:
- Actovegin 1200 mg: Actovegin 1200 mg, infusion, intravenously, once daily for up to 2 weeks followed by actovegin 200 mg, tablets, orally, thrice daily (1200 mg/day) for up to 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Actovegin 1200 mg | Total
Number analyzed (Participants) | 182 | 184 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (6.56) | 63.7 (6.76) | 63.3 (6.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 155 | 160 | 315
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 173 | 179 | 352
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 154 | 156 | 310
  Kazakhstan | 12 | 12 | 24
  Georgia | 16 | 16 | 32
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.0 (7.66) | 172.1 (7.43) | 172.1 (7.53)
Weight [Mean (Standard Deviation); unit: kilogram (Kg)] | 81.17 (12.483) | 81.30 (13.351) | 81.24 (12.909)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 27.42 (3.733) | 27.44 (4.131) | 27.43 (3.933)
PAD Stage II Duration [Mean (Standard Deviation); unit: years] | 5.482 (4.2019) | 5.283 (4.9374) | 5.382 (4.5812)
Diabetic Status [Count of Participants; unit: Participants]
  Diabetic | 29 | 40 | 69
  Non-diabetic | 153 | 144 | 297
Location of the Lesion [Count of Participants; unit: Participants]
  Aorto-iliac segment | 8 | 6 | 14
  Femoro-popliteal segment | 85 | 88 | 173
  Both segments | 89 | 90 | 179
Ankle Brachial Index (ABI) at Bilateral (BL) [Mean (Standard Deviation); unit: ratio] — The ABI assessment was performed by measuring the systolic blood pressure (sBP) from both brachial arteries, posterior tibial arteries, and both dorsalis pedis arteries. ABI was calculated as ankle sBP divided by brachial sBP. Ankle sBP was the higher of two systolic blood pressures from a lower limb. Brachial sBP was the higher of systolic blood pressures from both upper limbs.
  ratio | 0.580 (0.1511) | 0.589 (0.1564) | 0.584 (0.1536)
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 69 | 69 | 138
  Former smoker | 82 | 76 | 158
  Never-smoked. | 31 | 39 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Initial Claudication Distance (ICD) at Week 12
Description: ICD was the distance walked at the onset of claudication pain or pain-free walking distance. ICD was assessed using treadmill testing. A fixed load treadmill test was carried out at 3.0 kilometer per hour (km/h) with a 10 percent (%) grade.
Time Frame: Baseline up to Week 12
Population: The full analysis set (FAS) included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid post-baseline value for assessment of primary endpoint. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Actovegin 1200 mg
Number analyzed (Participants) | 180 | 177
percent change | 21.99 (9.286) | 51.17 (9.187)
Statistical Analysis 1: Comparison: Placebo vs Actovegin 1200 mg; Least squares means, p-values were obtained using a mixed model for repeated measures (MMRM) analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0041, MMRM; Least square mean difference = 29.19, 95% CI 2-sided [9.35 to 49.02], Standard Error of Mean 10.083

2. Secondary Outcome: Percent Change From Baseline in ICD at Weeks 2 and 24
Description: ICD was the distance walked at the onset of claudication pain or pain-free walking distance. ICD was assessed using treadmill testing. A fixed load treadmill test was carried out at 3.0 km/h with a 10% grade.
Time Frame: Baseline up to Weeks 2 and 24
Population: The FAS included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid post-baseline value for assessment of primary endpoint. Participants evaluable for this measure at given time point were included for the assessment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Actovegin 1200 mg
Number analyzed (Participants) | 182 | 180
percent change
  Week 2 | 6.58 (8.131) | 22.45 (7.981)
  Week 24: number analyzed (Participants) | 176 | 174
  Week 24 | 25.12 (10.665) | 60.63 (10.614)
Statistical Analysis 1: Comparison: Placebo vs Actovegin 1200 mg; Week 2: Least squares means, p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0431, MMRM; Least square mean difference = 15.86, 95% CI 2-sided [0.49 to 31.24], Standard Error of Mean 7.814
Statistical Analysis 2: Comparison: Placebo vs Actovegin 1200 mg; Week 24: Least squares means, p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0047, MMRM; Least square mean difference = 35.51, 95% CI 2-sided [10.96 to 60.05], Standard Error of Mean 12.480

3. Secondary Outcome: Absolute Change From Baseline in Absolute Claudication Distance (ACD) at Weeks 2, 12 and 24
Description: ACD was the distance at which claudication pain becomes so severe that the participant was forced to stop, also known as maximal walking distance. ACD was assessed using treadmill testing. A fixed load treadmill test was carried out at 3.0 km/h with a 10% grade. The investigator will record the distance from walking start to the point where the participant is unable to walk anymore.
Time Frame: Baseline, Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Placebo | Actovegin 1200 mg
Number analyzed (Participants) | 182 | 180
meter
  Baseline | 134.5 (58.84) | 137.1 (72.76)
  Change at Week 2 | 17.61 (30.781) | 46.28 (179.356)
  Change at Week 12: number analyzed (Participants) | 180 | 177
  Change at Week 12 | 30.05 (50.530) | 75.51 (190.808)
  Change at Week 24: number analyzed (Participants) | 176 | 174
  Change at Week 24 | 36.37 (71.834) | 86.47 (227.491)
Statistical Analysis 1: Comparison: Placebo vs Actovegin 1200 mg; Week 2: p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0227, MMRM
Statistical Analysis 2: Comparison: Placebo vs Actovegin 1200 mg; Week 12: p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0007, MMRM
Statistical Analysis 3: Comparison: Placebo vs Actovegin 1200 mg; Week 24: p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0023, MMRM

4. Secondary Outcome: Percentage of Participants With Rest Pain at Weeks 12 and 24
Description: Rest pain was defined as a continuous burning pain, that begins, or is aggravated, after reclining or elevating the limb and is relieved by sitting or standing.
Time Frame: Weeks 12 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Actovegin 1200 mg
Number analyzed (Participants) | 182 | 180
percentage of participants
  Week 12 | 0 | 0.6
  Week 24: number analyzed (Participants) | 180 | 176
  Week 24 | 1.1 | 0.6
Statistical Analysis 1: Comparison: Placebo vs Actovegin 1200 mg; Week 12; Test type: Non-Inferiority — As the sample size was too small, clinically significant difference in actovegin and placebo could not be defined, the non-inferiority margin was defined as priori based on clinical reasoning; p = 0.9592, Regression, Logistic — p-values were obtained using logistic regression adjusting for treatment
Statistical Analysis 2: Comparison: Placebo vs Actovegin 1200 mg; Week 24; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.5823, Regression, Logistic — p-values were obtained using logistic regression adjusting for treatment

5. Secondary Outcome: Percentage of Participants With Revascularization Procedures at Week 24
Description: Revascularization was defined by a Thrombolysis in Myocardial Infarction (TIMI) score of 2 or 3 following use of the Penumbra System. TIMI scores were used to describe blood flow at the treated vessel with 0 designating no flow and 3 for normal flow.
Time Frame: Week 24
Population: The FAS included all participants who were randomized, received at least 1 dose of study drug, and had at least 1 valid post-baseline value for assessment of primary endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Actovegin 1200 mg
Number analyzed (Participants) | 182 | 180
percentage of participants | 0.0 | 1.1
Statistical Analysis 1: Comparison: Placebo vs Actovegin 1200 mg; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.9424, Regression, Logistic — p-values were obtained using logistic regression adjusting for treatment

6. Secondary Outcome: Change From Baseline in 36-Item Short Form Survey (SF-36) at Weeks 12 and 24
Description: The SF-36 was a questionnaire that evaluated a participant's health related quality of life. SF-36 included 36 questions related to 8 health dimensions: physical functioning, role-physical (role limitations due to physical health problems), bodily pain, general health, vitality (energy/fatigue), social functioning, role-emotional (role limitations due to emotional problems), and mental health. Based on these 4 scales (physical functioning, role-physical, bodily pain, general health), the physical health score was generated which ranges between 0 and 100, with higher scores indicating a better quality of life. Based on these 4 scales (vitality, social functioning, role-emotional, and mental health), the mental health score was generated which ranges between 0 and 100, with higher scores indicating a better quality of life.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Actovegin 1200 mg
Number analyzed (Participants) | 182 | 180
points on a scale
  Physical Health Score: Baseline | 39.533 (6.3023) | 39.905 (6.5138)
  Physical Health Score: Change at Week 12: number analyzed (Participants) | 180 | 177
  Physical Health Score: Change at Week 12 | 2.029 (5.1633) | 2.368 (5.3725)
  Physical Health Score: Change at Week 24: number analyzed (Participants) | 177 | 176
  Physical Health Score: Change at Week 24 | 1.752 (6.1229) | 2.333 (5.1950)
  Mental Health Score: Baseline | 47.961 (9.4891) | 47.531 (9.8667)
  Mental Health Score: Change at Week 12: number analyzed (Participants) | 180 | 177
  Mental Health Score: Change at Week 12 | 1.134 (7.2459) | 2.434 (8.2234)
  Mental Health Score: Change at Week 24: number analyzed (Participants) | 177 | 176
  Mental Health Score: Change at Week 24 | 0.571 (8.6698) | 3.063 (9.0286)
Statistical Analysis 1: Comparison: Placebo vs Actovegin 1200 mg; Physical Health Score: Week 12; Least squares means, p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.3758, MMRM
Statistical Analysis 2: Comparison: Placebo vs Actovegin 1200 mg; Physical Health Score: Week 24; Least squares means, p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.1412, MMRM
Statistical Analysis 3: Comparison: Placebo vs Actovegin 1200 mg; Mental Health Score: Week 12; Least squares means, p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.1009, MMRM
Statistical Analysis 4: Comparison: Placebo vs Actovegin 1200 mg; Mental Health Score: Week 24; Least squares means, p-values were obtained using a MMRM analysis of covariance with treatment, center, sex, age group, smoking status, diabetic status, visit and treatment-by-visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0015, MMRM

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are adverse events that started after the first dose of study drug up to Day 168
Description: At each visit the investigator had to assess any occurrence of adverse events. Participants may report adverse events occurring at any other time during the study. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Actovegin 1200 mg
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/184
Serious Adverse Events (participants affected / at risk) | 3/182 | 9/184
Other Adverse Events (participants affected / at risk) | 20/182 | 23/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=182) | Actovegin 1200 mg (N=184)
Angina unstable (Cardiac disorders) | 0 | 1
Gangrene (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=182) | Actovegin 1200 mg (N=184)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Carbohydrate metabolism disorder (Congenital, familial and genetic disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 5
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Chronic hepatitis C (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03469349/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03469349/SAP_001.pdf